CLINICAL TRIAL: NCT06594861
Title: Follow-up of Clinical Manifestations and Inflammation-related Parameters in Individuals with Autoantibodies Against Ro/SSA and La/SSB
Brief Title: Follow-up Study of Individuals with Autoantibodies Against Ro/SSA and La/SSB
Acronym: ProgreSS
Status: Recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Albin Björk, Principal Investigator, Karolinska Institutet
Other Study IDs: 2023-04569-01
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Autoantibodies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Sampling includes tubes for serum, plasma, RNA and DNA extraction, as well as for cell separation.
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (2):
- Individuals with autoantibodies against Ro/SSA and/or La/SSB
  Interventions: Other: No intervention
- Individuals without autoantibodies against Ro/SSA and/or La/SSB
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention.

SUMMARY:
In this study, individuals with autoantibodies against Ro/SSA and La/SSB will be followed with regard to clinical manifestations and immunological parameters to identify immunological changes, environmental factors, and early clinical symptoms that characterize the progression from serological autoreactivity to clinically manifest disease.

DETAILED DESCRIPTION:
Autoimmune diseases are a diverse group of conditions characterized by chronic inflammation and tissue damage. In systemic autoimmune diseases such as Sjögren disease and systemic lupus erythematosus (SLE), two specific types of autoantibodies targeting the bodys own proteins, Ro/SSA and La/SSB, are often present.

It is well known that some individuals with autoantibodies against Ro/SSA and/or La/SSB never develop any systemic rheumatic disease, while in others, the presence of these autoantibodies is a sign of impending disease. The condition of so-called serological autoreactivity, which can persist for decades, and how clinical disease subsequently develops is very little studied. There is currently a lack of knowledge regarding the environmental factors that contribute to the emergence of autoantibodies against Ro/SSA and/or La/SSB and the immunological mechanisms that lead to disease development in some individuals but not in others.

This project aims to enhance the understanding of the condition of serological autoreactivity against Ro/SSA and La/SSB. The specific goal is to identify immunological changes, environmental factors, and early clinical symptoms that characterize the progression from serological autoreactivity to clinically apparent disease. Understanding the immunological mechanisms that trigger the transition to disease is crucial for enabling earlier diagnosis and treatment, as well as for better comprehending the fundamental mechanisms underlying the development of autoimmune disease.

This will be achieved by:

1. Clinically characterizing at-risk individuals who carry autoantibodies against Ro/SSA and/or La/SSB through medical consultations at a rheumatology specialist clinic.
2. Immunologically characterizing at-risk individuals in comparison with healthy individuals through blood sampling and immunological analyses.
3. Collecting data on exposure to environmental and lifestyle factors that could potentially increase the risk of autoimmunity.

Study participants are offered annual follow-up assessments for four years after the inclusion visit (i.e., a total of 4 study visits per participant). Participants that develop new symptoms during the study are be offered additional medical visits for assessment. At the final follow-up visit, participants will be asked for their consent to be contacted by phone to inquire about any new symptoms and to schedule new blood tests after two and five years, respectively.

ELIGIBILITY:
Inclusion Criteria:

To be included in the risk group, the following criteria must be met:

- At least one instance of testing positive for Ro/SSA or La/SSB, regardless of the method used.

To be included in the control group, the individual must:

- Have no rheumatologic disease and no autoantibodies against Ro/SSA or La/SSB.

Exclusion Criteria:

1. Below 18 years of age
2. Inability to consent to their own participation
3. Ongoing infection or severe illness where the study physician deems participation in the study not to be in the individuals best interest
4. Inability to read and understand Swedish, and therefore unable to complete the forms and questionnaires included in the project

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals who have been evaluated at a rheumatology specialist clinic or followed by a pediatric cardiologist due to autoantibodies against Ro/SSA and/or La/SSB are invited to participate in the study. Healthy controls are invited through advertisements.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-02-09 (Actual); Primary Completion 2038-12 (Estimated); Study Completion 2038-12 (Estimated)

PRIMARY OUTCOMES:
Development of a rheumatic disease | From enrolment to a maximum of 9 years of follow-up.
  The number of participants that develop rheumatic disease among the individuals with autoantibodies will be assessed

SECONDARY OUTCOMES:
Frequency of clinical symptoms | From enrolment to a maximum of 9 years of follow-up.
  The frequencies of clinical signs and symtoms thought to be related to anti-SSA/Ro and anti-SSB/La autoantibodies will be assessed

CONTACTS AND LOCATIONS:
Locations (1):
- Centrum för reumatologi, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No